CLINICAL TRIAL: NCT02117674
Title: Full Spectrum vs. Standard Forward-viewing Colonoscopy With and Without Right-colon Retroflexion: a Randomized, Bicentric Back-to-back Study
Brief Title: Full Spectrum vs. Standard Forward-viewing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, ATHANASIOS SIOULAS, Dr, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FUSE-001
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Colon Neoplasms
Keywords: colonoscopy; adenoma detection rate; full spectrum colonoscopy; right colon retroflexion; feasibility
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard forward-viewing colonoscopy (Active Comparator): polyp detection with standard forward-viewing colonoscopy polyp detection in the right colon with scope retroflexion
  Interventions: Procedure: standard forward-viewing colonoscopy; Procedure: full-spectrum colonoscopy; Procedure: right colon retroflexion
- full-spectrum colonoscopy (Active Comparator): polyp detection with full-spectrum colonoscopy polyp detection in the right colon with scope retroflexion
  Interventions: Procedure: standard forward-viewing colonoscopy; Procedure: full-spectrum colonoscopy; Procedure: right colon retroflexion

INTERVENTIONS:
Procedure: standard forward-viewing colonoscopy — examination of the colon with a conventional colonoscope
  Other Names: conventional colonoscopy
Procedure: full-spectrum colonoscopy — examination of the colon with full-spectrum colonoscope
  Other Names: fuse endoscopy
Procedure: right colon retroflexion — examination of the right colon with scope retroflexion (both with conventional and fuse scope)
  Other Names: retroflexion

SUMMARY:
The aim of this study is to evaluate FUSE-colonoscopy in terms of feasibility and its possible additive contribution in the detection of important lesions, namely polyps and cancers, compared to the standard "forward-viewing" approach, with and without the addition of the right-colon retroflexion technique, in a series of patients undergoing back-to-back screening or surveillance colonoscopies in a randomized fashion.

DETAILED DESCRIPTION:
We changed the anticipated number of subjects enrollment for study: NCT02117674 from 120 to 200 based on the following sample size estimation:

Tandem colonoscopies studies results, show that novel endoscopic technologies detect about 20% more adenomas than those conventional colonoscopy does (missed adenomas). Since FUSE colonoscopy cannot be considered as a perfect examination, we hypothesize that conventional colonoscopy will detect one third of the missed adenomas that FUSE detects in a similar setting. Therefore a sample size of 120 adenomas achieves 80% power to detect an odds ratio of 3.0 using a two-sided McNemar test with a significance level of 0.05. The odds ratio is equivalent to a difference between two paired proportions of 14% which occurs when the proportion of detected missed adenomas during FUSE is 21% and the proportion of missed adenomas during conventional colonoscopy is 7%. During one year period before the study initiation, our colonoscopy performance quality data show that we detect a mean number of adenomas per patient equal of 0.7 in a population similar to the one recruited in our study. Therefore, 172 patients overall will be required to detect 120 adenomas. Given the uncertainty of our estimation and in order to cope with patients exclusions, withdrawals and unexpected incomplete colonoscopies, we decided to recruit 200 patients.

A more extensive description regarding the investigators study is provided in the following fields.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing elective screening or surveillance colonoscopy
* symptomatic adults with indication for colonoscopy

Exclusion Criteria:

* age over 80 years
* poor overall health (ASA III, IV)
* recent abdominal surgery
* presence of abdominal wall hernias
* active colitis
* multiple right colon diverticula
* previous bowel resection
* inflammatory bowel disease
* polyposis syndromes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
polyp detection rate | one week
  per colon segment and for the entire colon

SECONDARY OUTCOMES:
colonoscopy completion | one week
  colonoscopy completion rate
procedure time | one week
  intubation and withdrawal time
adverse events | one week
  adverse events rate
endoscopist's satisfaction | one week
  endoscopist's satisfaction quantified using a scale from 0 (not satisfied) to 10 (completely satisfied)
feasibility of the retroflexion in the right colon by trainee | one week
  feasibility of retroflexion in the right colon by trainee, meaning if the trainee managed to perform the right colon retroflexion or not
feasibility of retroflexion in the right colon by the consultant | one week
  feasibility of retroflexion in the right colon by the consultant, meaning if the consultant managed to perform the right colon retroflexion or not
patients' satisfaction | one week
  patients' satisfaction, quantified using a scale from 0 (not satisfied at all) to 10 (completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: KONSTANTINOS TRIANTAFYLLOU, Prof, Study Director — Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Unit, Attikon University General Hospital, University of Athens, Greece; GEORGE ALEXANDRAKIS, Dr, Study Director — 417 NIMTS VETERANS HOSPITAL
Locations (2):
- Greece (2):
  - 417 Nimts Veterans Hopsital, Athens
  - Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Unit, Attikon University General Hospital, Athens

REFERENCES:
- [Background] Hewett DG, Rex DK. Miss rate of right-sided colon examination during colonoscopy defined by retroflexion: an observational study. Gastrointest Endosc. 2011 Aug;74(2):246-52. doi: 10.1016/j.gie.2011.04.005. Epub 2011 Jun 15. PMID 21679946
- [Background] Gralnek IM, Segol O, Suissa A, Siersema PD, Carr-Locke DL, Halpern Z, Santo E, Domanov S. A prospective cohort study evaluating a novel colonoscopy platform featuring full-spectrum endoscopy. Endoscopy. 2013 Sep;45(9):697-702. doi: 10.1055/s-0033-1344395. Epub 2013 Aug 12. PMID 23939509
- [Derived] Papanikolaou IS, Apostolopoulos P, Tziatzios G, Vlachou E, Sioulas AD, Polymeros D, Karameris A, Panayiotides I, Alexandrakis G, Dimitriadis GD, Triantafyllou K. Lower adenoma miss rate with FUSE vs. conventional colonoscopy with proximal retroflexion: a randomized back-to-back trial. Endoscopy. 2017 May;49(5):468-475. doi: 10.1055/s-0042-124415. Epub 2017 Jan 20. PMID 28107765